CLINICAL TRIAL: NCT02474121
Title: MarrOwStim™ PAD Kit for the Treatment of Critical LimB IschemIa (CLI) in Subjects With Severe Peripheral ArteriaL DiseasE (PAD) (MOBILE) - Continued Access
Brief Title: Safety and Efficacy of Autologous Concentrated Bone Marrow Aspirate for Critical Limb Ischemia - Continued Access
Acronym: MOBILE-CA
Status: No longer available | Type: Expanded Access
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: BB-IDE 13996 (CA)
Record Dates: First submitted 2015-06-15; First posted 2015-06-17 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Peripheral Arterial Disease; Peripheral Vascular Diseases; Critical Limb Ischemia
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia

INTERVENTIONS:
Device: Bone marrow concentration device — Collection of autologous bone marrow aspirate and point-of-care concentration using the bone marrow concentration device, followed by intramuscular injection of concentrated bone marrow aspirate (cBMA) into the affected limb
  Other Names: MarrowStim™ PAD Kit; Bone Marrow Concentrate; Bone Marrow Mononuclear Cells

SUMMARY:
This study will continue to evaluate the performance of the MarrowStim™ PAD Kit to treat subjects with critical limb ischemia (CLI) caused by severe PAD.

DETAILED DESCRIPTION:
This is a continued access enrollment intended for subjects with critical limb ischemia (CLI) that are unsuitable for revascularization. The investigational treatment utilizes autologous concentrated bone marrow aspirate (cBMA) at the point of care. The bone marrow aspirate is obtained from the subject's hip, concentrated with a bone marrow concentration device, and delivered intramuscularly to the affected limb. Subjects meeting the inclusion/exclusion criteria will be treated with the MarrowStim™ PAD Kit and followed for a total of five years. Information on subject outcomes, such as the occurrence of amputation and death, as well as measurements of rest pain, blood flow (ankle-brachial index, toe-brachial index), and quality of life will be collected. Safety information (via adverse event reporting) will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral lower extremity ischemia due to advanced peripheral arterial disease
* Unsuitable for revascularization
* Minor tissue loss (Rutherford Category 5) or ischemic rest pain (Rutherford Category 4)
* Competent to give consent
* No current malignancy or history of previous malignancy within the last five years, with the exception of adequately treated non-melanoma skin cancer (evidence of standard preventative cancer screenings required)

Exclusion Criteria:

* Major tissue loss (Rutherford Category 6)
* Diabetics with uncontrolled or untreated proliferative retinopathy
* Poorly controlled diabetes mellitus with HbA1C > 10%
* Uncompensated congestive heart failure and/or other conditions that preclude general anesthesia
* Myocardial infarction or stroke within last 90 days
* Elevated liver function tests (AST or ALT more than twice the upper limit of normal)
* Renal disease (creatinine > 2.5 mg/dl) or chronic hemodialysis
* White blood cell count < 3,000/µL or > 15,000/µL, platelet count < 100,000/µL, or hematocrit < 32%
* Topical growth hormone therapy within last 90 days, or injected growth hormone therapy within last 180 days
* Disease of central nervous system and/or other conditions that impair cognitive function
* Two or more episodes of pulmonary embolus with a documented DVT in index leg or history of DVT in index leg without evidence of clot resolution
* Current infection of index leg
* Pregnant women (negative urine pregnancy test required)
* Lower extremity venous disease with pitting edema in index leg
* Recent history (in the 6 months prior to screening) of bone marrow disease or treatment with any medication or procedure which adversely affects the bone marrow and would prohibit transplantation
* Current osteomyelitis in index leg
* Existing HIV diagnosis
* Organ transplant recipients
* Known terminal disease process with life expectancy less than one year
* Severe concomitant disease(s) or any additional condition(s) which the investigator feels constitute(s) criteria for exclusion of a particular subject
* Major amputation required within 30 days
* Inclusion in any other clinical study that may affect the outcome of this study
* Uncorrected stenosis(es) of greater than 50% in the common and/or external iliac artery and/or common femoral artery of the index leg.

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - Piedmont Hospital, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - Holy Name Medical Center, Teaneck, New Jersey
  - The Mount Sinai Hospital, New York, New York
  - Weill Cornell Medical College/New York Presbyterian Hospital, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Murphy MP, Lawson JH, Rapp BM, Dalsing MC, Klein J, Wilson MG, Hutchins GD, March KL. Autologous bone marrow mononuclear cell therapy is safe and promotes amputation-free survival in patients with critical limb ischemia. J Vasc Surg. 2011 Jun;53(6):1565-74.e1. doi: 10.1016/j.jvs.2011.01.074. Epub 2011 Apr 22. PMID 21514773
- [Derived] Wang SK, Green LA, Gutwein AR, Drucker NA, Babbey CM, Gupta AK, Fajardo A, Motaganahalli RL, Wilson MG, Murphy MP. Ethnic minorities with critical limb ischemia derive equal amputation risk reduction from autologous cell therapy compared with whites. J Vasc Surg. 2018 Aug;68(2):560-566. doi: 10.1016/j.jvs.2017.11.088. Epub 2018 Mar 1. PMID 29503004